CLINICAL TRIAL: NCT01178840
Title: A Randomized Cross-Over Study of Vaginal Semen Exposure and Clinical Failure Comparing the PATH Woman's Condom and the FC2 Female Condom
Brief Title: Prostate Specific Antigen (PSA) and Acute Failure Modes Study of the PATH Woman's Condom and FC2 Female Condom
Acronym: CONRAD-108
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CONRAD-108
Record Dates: First submitted 2010-08-04; First posted 2010-08-10 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2012-03

CONDITIONS: Birth Control
Keywords: female condom; condom; clinical failure; prostate-specific antigen; semen exposure; acceptability; Prevention of semen exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WC then FC2 (Other): The couples will use 4 PATH Woman's Condom then 4 FC2 female condom.
  Interventions: Device: WC then FC2
- FC2 then WC (Other): The couples will use 4 FC2 female condom then 4 PATH Woman's Condom.
  Interventions: Device: FC2 then WC

INTERVENTIONS:
Device: WC then FC2 — 4 uses of WC followed by 4 uses of FC2
  Other Names: WC = Woman's Condom; FC2 = Female Condom 2
  Arms: WC then FC2
Device: FC2 then WC — 4 uses of WC followed by 4 uses of FC2
  Other Names: WC = Woman's Condom; FC2 = Female Condom 2
  Arms: FC2 then WC

SUMMARY:
This is a comparative, open-label two-period crossover study of up to 505 couples comparing the PATH Woman's Condom to the FC2 female condom. California Family Health Council will enroll up to 505 couples to have 375 complete both periods. The study will provide data on functional performance, vaginal semen exposure, safety, and acceptability of the two female condoms.

Both partners will be required to come to the clinic to be consented for the study. If both members of the couple meet all eligibility requirements, they will each sign an informed consent form and will be enrolled as a couple. The couples will be randomized to one of two female condom use sequences for the two periods (WC then FC2 or FC2 then WC). For the first period of 2-4 weeks, the couple will be asked to have sex once without a condom and 4 times using the first assigned female condom. For the second period of 2-4 weeks, the couple will be asked to have sex 4 times using the second assigned female condom. In the first period, the couple will have one act of unprotected sex for which they will collect pre- and post-coital vaginal swabs. The couple will also use 4 female condoms of the assigned type. They will be asked to collect pre- and post-coital vaginal swabs and a post-coital swab from the condom interior. The couple will complete a detailed Condom Use Questionnaire together after each condom use. An Acceptability Questionnaire will be completed separately by males and females at the end of each study period. Couples may have additional acts of sex during each period as they desire but will not have sex at least 48 hours prior to each study sex act. After a follow-up visit, the procedures will be repeated with 4 of the second assigned condom type but without the collection of vaginal swabs at unprotected intercourse. Each couple will be enrolled for about 2-3 months, depending on the intervals between sex acts. Clinicians evaluating product-relatedness of AEs will be blinded to the condom type used. Male partners will be requested to attend the final visit, and, if they experience adverse events, the followup and/or unscheduled visits.

DETAILED DESCRIPTION:
Purpose: To compare the performance of a new female condom (PATH Woman's Condom) with an FDA-approved female condom (FC2), as assessed by reported clinical failure and vaginal PSA

Design: This is a comparative, open-label two-period crossover study of up to 505 couples comparing the PATH Woman's Condom to the FC2 female condom. We will enroll up to 505 couples at the California Family Health Council to have 375 complete both periods. The study will provide data on functional performance, vaginal semen exposure, safety, and acceptability of the two female condoms.

Primary objective: To compare the performance of the PATH Woman's Condom (WC) to the FC2, as assessed by self-reported total clinical failure and its components (clinical breakage, slippage, misdirection, and invagination).

Secondary objectives:

* To compare the ability of the WC and the FC2 to prevent vaginal exposure to semen, as indicated by detection of PSA within the vagina
* To calculate the sensitivity and specificity of reported failures using PSA as the gold standard for the presence of semen
* To compare acceptability of the WC and FC2

Study Population: Healthy heterosexual couples at least 18 years of age and at low risk for pregnancy or STIs.

Study Size: up to 505 couples divided between multiple recruitment locations under one center.

Study Duration: Accrual will require approximately 14 months. Each couple will be expected to complete the study in 2-3 months. Therefore, the clinical portion of the study should be completed within approximately 17 months. Data preparation, analysis, and report writing are expected to require up to 7 months after completion of the clinical portion.

Treatment Regimen: The couples will be randomized to one of two condom use sequences (WC then FC2 or FC2 then WC). Four condoms of each type will be used by couples over two 2-4 week periods. For first period, one set of pre- and post-coital vaginal swabs will be collected around unprotected intercourse. For each coital act where a condom is used in the period, pre and post-coital vaginal swabs and a post-coital condom swab will be collected. A Condom Use Questionnaire will be completed after each condom use. An Acceptability Questionnaire will be completed at the end of each period. After a follow-up visit, these procedures will be repeated with the second 4 condoms, without collection of vaginal swabs at unprotected intercourse.

Study Center: California Family Health Council

Funding Source: United States Agency for International Development (USAID) & National Institute for Child Health and Development (NICHD)

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual couples
* Mutual monogamy for 3 or more months
* Both partners are 18 years of age or greater
* Using effective contraception for more than 3 months, including hormonal methods (oral, injectable, or transdermal), intrauterine device, contraceptive implant, male or female sterilization
* Agree to remain monogamous for the duration of the study
* Agree not to wear any genital piercing jewelry while using study condoms
* Agree not to use sex toys or drugs intended to enhance or diminish sexual response when using a study condom
* Evidence of general good health without contraindication to sexual activity
* Couple has vaginal intercourse at least 4 times in a typical month
* Male partner agrees to ejaculate during intercourse using female condoms
* Willing and able to participate as required by protocol

Exclusion Criteria:

Exclusion criteria for couple (either partner)

* Intent or desire to become pregnant within 3 months
* STIs in the past 6 months, including chlamydia, gonorrhea, trichomoniasis, syphilis, or newly acquired HSV
* Couple routinely uses condoms due to concern for STIs (for more than 90% of sex acts)
* Known HIV infection
* At high risk for HIV infection, including having shared injection drug needles or having had sex with someone suspected to have HIV (without having had a negative HIV test since the possible exposure).
* Allergies to polyurethane or nitrile plastics, or vaginal lubricants (silicone or Astroglide)
* Recent surgery or biopsy of the male or female genitalia, within the past 60 days including the vulva, vagina, cervix, penis, prostate, vas deferens, or testes
* Current participation in a study or other research involving a drug, device, or other product. (Participation in an observational study is not exclusionary).

Exclusion criteria for female partner

* Positive pregnancy test
* Within 2 months of the end of pregnancy
* Concern for current pregnancy: history of unprotected intercourse since last menses without consistent use of other contraception
* Use of a contraceptive vaginal ring (Nuvaring)
* Current use of vaginal products, for treatment of vaginal infection
* Routine use of diaphragm or vaginal pessary
* Polycystic ovarian syndrome (oligomenorrhea and hirsutism or prior diagnosis)
* Distorted vaginal anatomy (e.g. vaginal septum or pelvic prolapse)

Exclusion criteria for male partner

* Difficulty maintaining an erection or achieving ejaculation in the last two months
* At high risk for HIV infection, including having had anal sex with a man in the last year
* Prior prostate surgery
* History of or current prostate cancer
* Use of medication for a prostate condition
* Hypospadias or other abnormal penile or male urethral anatomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 505 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Self-reported clinical failure including clinical breakage, misdirection, slippage, and invagination | 8 condom uses over up to 3 months

SECONDARY OUTCOMES:
Vaginal PSA levels | 8 condom uses over up to 3 months
  For each sex act, the change in vaginal PSA will be examine. The change in PSA will be equal to the PSA value from the POST-coital swab minus the PSA value from the PRE-coital swab. We will also collect swabs from one sex act without a condom as a positive control.
Female condom acceptability | 8 condom uses over up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jill L Schwartz, MD, Study Director — CONRAD
Locations (1):
- California Family Health Council, Los Angeles, California, United States

REFERENCES:
- [Derived] Walsh TL, Snead MC, St Claire BJ, Schwartz JL, Mauck CK, Frezieres RG, Blithe DL, Archer DF, Barnhart KT, Jensen JT, Nelson AL, Thomas MA, Wan LS, Weaver MA. Comparison of self-reported female condom failure and biomarker-confirmed semen exposure. Contraception. 2019 Nov;100(5):406-412. doi: 10.1016/j.contraception.2019.07.143. Epub 2019 Aug 2. PMID 31381878